CLINICAL TRIAL: NCT04406181
Title: Effect on the COVID-19 Pandemic-induced Reduction in Elective Surgery on Medical Events and Psychological Well-being of Patients Waiting for Cardiac Surgery
Brief Title: Psychological Well-being of Patients Awaiting for Cardiac Surgery During the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID-19 Cardiac psy wellbeing
Record Dates: First submitted 2020-04-28; First posted 2020-05-28 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Anxiety and Fear; Anxiety Depression; Anxiety Postoperative; Psychological Stress
Keywords: cardiac surgery; postoperative consultation; postponed elective surgery; COVID-19
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological; COVID-19 | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- operation deferred (Other): Adult patients whose operation date has been deferred due to the pandemic
  Interventions: Behavioral: HADS; Behavioral: a survey
- no operation date (Other): Patients who did not have had an operation date and who were told to need cardiac surgery before the pandemic started
  Interventions: Behavioral: HADS; Behavioral: a survey
- postoperative consultation deferred (Other): Patients who have been operating on during the month before the pandemic
  Interventions: Behavioral: HADS; Behavioral: a survey

INTERVENTIONS:
Behavioral: HADS — Hospital Anxiety and Depression Scale
  Other Names: questionnaire
Behavioral: a survey — made up specifically for issues concerning the medical/psychological/access aspects during the COVID-19 outbreak

SUMMARY:
The effect and impact of postponing cardiac surgery / creating a waiting list as a result of COVID-19 on patients, both psychologically and symptomatically on three groups of patients:

1. The degree of anxiety and/or depression induced by their altered medical care trajectory.
2. The incidence of medical problems induced by deferred elective surgery or delayed postoperative ambulatory visit
3. The occurrence of reduced access to medical and psychological help

DETAILED DESCRIPTION:
A prospective study by means of a questionnaire, specifically designed for each of the three groups.

1. Adult patients whose operation date has been deferred
2. Patients who did not have had an operation date
3. Patients who have been operating on during the month before

Each group will receive a twofold questionnaire:

Part I: Hospital Anxiety and Depression Scale (HADS), a robust questionnaire used for hospitalized and non-hospitalized patients gauging the degree of anxiety and/or depression, irrespective of their specific medical condition. All three groups receive the same list of questions.

-Part II: a questionnaire made up specifically for issues concerning the medical/psychological/access aspects during the COVID-19 outbreak. Each of the three groups will receive a questionnaire, adapted to the group they are assigned to.

The questionnaires will be delivered by the use of Qualtrics or on paper. Timing and mode of presentation (Qualtrics or fill-in paper on admission) of the questionnaire will depend on the length of the quarantine measures.

ELIGIBILITY:
Inclusion Criteria:

All adult patients whose operation date has been deferred due to the pandemic COVID-19.

All patients who did not have had an operation date before the pandemic COVID-19.

All patients who have been operating on during the month before the pandemic COVID-19.

Exclusion Criteria:

N/A

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety/depression by means of Hospital Anxiety and Depression Scale (HADS) | 10 minutes
  The degree of anxiety and/or depression in all three groups, induced by their altered medical care trajectory. 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Medical problems induced by deferred elective surgery or delayed postoperative ambulatory visit | 10 minutes
  The incidence of medical problems induced by deferred elective surgery or delayed postoperative ambulatory visit by means of an adjusted survey.
Reduced access to medical and psychological help | 10 minutes
  The occurrence of reduced access to medical and psychological help by means of an adjusted survey.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nijs, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Mark La Meir, Phd, MD, Study Director — Universitair Ziekenhuis Brussel; Ashley Welch, MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium